CLINICAL TRIAL: NCT05951322
Title: The Influence of Extra Corporeal Shock Wave Versus Phonophoresis on Pain Severity and Functional Disability in Patients With Sub Acromial Impingement Syndrome. A Randomized Clinical Trial.
Brief Title: Extra Corporeal Shock Wave Versus Phonophoresis in Sub Acromial Impingement Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Principal Investigator, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECM#2023-1102
Record Dates: First submitted 2023-06-09; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sub Acromial Impingement Syndrome
Keywords: Extra corporeal shock wave; phonophoresis; sub acromial impingement syndrome
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Phonophoresis

STUDY DESIGN:
Intervention Model Description: Participants were identified and recruited over 5-month period. Thirty-six patients diagnosed clinically with shoulder impingement syndrome (according to location of trigger points at rotator cuff muscles and aggravation of pain with overhead activities) were randomly assigned in two groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome asseser is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave therapy (Experimental): All patients were received (ESWT) at sitting position, exposed the affected shoulder, the shoulder adducted and elbow extended and the shock wave applicator was directed in most tender point near the insertion of rotator cuff at greater tuberosity under the acromion [23].
  The treatment area was prepared with a coupling gel to minimize the loss of shockwave at the interface between applicator tip and skin.
  Each patient was received (6000 shocks,21000 shock/ session, 3 session 2 weeks apart, energy flux density 0.22 mJ/mm2, energy level 5-7, pulse rate 160/min., 2-3Hz)
  Interventions: Device: Shockwave therapy
- Phonophoresis (Active Comparator): Pagani ultrasound apparatus 200 cosistts of multi frequency head(1 and 3 MHz), surface area 4 cm², continuous and pulsed mode, main voltages: 100-240-VAC.50/60Hz.
  Interventions: Device: Phonophoresis

INTERVENTIONS:
Device: Shockwave therapy — Radial extracorporeal shock wave device, it is serial number (1107394), medispec and connected to electrical supply 115/220 A C frequency.
  Arms: Shockwave therapy
Device: Phonophoresis — Pagani ultrasound apparatus 200 cosistts of multi frequency head(1 and 3 MHz), surface area 4 cm², continuous and pulsed mode, main voltages: 100-240-VAC.50/60Hz.
  Arms: Phonophoresis

SUMMARY:
shoulder sub acromial impingement syndrome is an encroachment of subacrormial tissues, rotator cuff, subacrormial bursa, and the long head of the biceps tendon, as a result of narrowing of the subacrormial space. Activities requiring repetitive or sustained use of the arms over head often predispose the rotator cuff tendon to injury. Hence the objective of the study is to examine the influence of extra corporeal Shock wave versus phonophoresis on pain severity and functional disability in patients with sub acromial impingement syndrome.

DETAILED DESCRIPTION:
Background: shoulder sub acromial impingement syndrome is an encroachment of subacrormial tissues, rotator cuff, subacrormial bursa, and the long head of the biceps tendon, as a result of narrowing of the subacrormial space. Activities requiring repetitive or sustained use of the arms over head often predispose the rotator cuff tendon to injury. Objective of the study: To examine the influence of extra corporeal Shock wave versus phonophoresis on pain severity and functional disability in patients with sub acromial impingement syndrome. Subjects and Methods: Thirty patients diagnosed as shoulder impingement syndrome stage II Neer classification due to mechanical causes. Patients were randomly distributed into two equal groups. The first group consisted of 15 patients with a mean age of 45.46 (+ 8.64) received therapeutic exercises( stretching exercise of posterior shoulder capsule and strengthening exercises of shoulder muscles) and shockwave therapy (6000 shock, 2000/session, 3 sessions, 2 weeks a part, 0.22mJ/mm2) years. The second group consisted of 15 patients with a mean age of 46.26 (+ 8.05) received same therapeutic exercises and phonophoresis (3 times per week, each other day, for 4 consecutive weeks). Patients were evaluated pretreatment and post treatment for shoulder pain severity, shoulder functional disability, shoulder flexion, abduction and internal rotation motions.

ELIGIBILITY:
Inclusion Criteria:

* The patient reported a positive "Neer sign" and" Hawkins sign".
* The patient reported pain with active shoulder elevation in the scapular plane (eg: welders, plate workers, slaughterhouse workers and over head playing athletes).
* The patient reported pain with palpation of the rotator cuff tendons.
* The patient reported pain with resisted isometric abduction.

Exclusion Criteria:

* Frozen shoulder.
* Rotator cuff tear.
* Glenohumeral or acromioclavicular arthritis.
* Implented pace maker.
* Pregnancy

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Pain assessed by (Visual analog scale (VAS). VAS is a scale that allows continuous data analysis and uses a 10cm line with 0 (no pain) and 10 (worst pain) on the other end .Patients were asked to place a mark a long the line to denote their level of pain.
Pain intensity | 6 weeks
  Pain assessed by (Visual analog scale (VAS). VAS is a scale that allows continuous data analysis and uses a 10cm line with 0 (no pain) and 10 (worst pain) on the other end .Patients were asked to place a mark a long the line to denote their level of pain.

SECONDARY OUTCOMES:
Functional disability | Baseline
  It was assessed by using the shoulder pain and disability index (SPADI) which is a valid and reliable index for measuring shoulder pain and disability. It consists of two parts, part one which assesses pain and part two which assesses functional disability. Scores were calculated as follow, in part one pain scores in all questions were added, and the mean value was chosen. In part two functional score of all questions were added and the mean value was chosen for the purpose of data analysis. Final score for each part was statistically analyzed separately.
Functional disability | 6 weeks
  It was assessed by using the shoulder pain and disability index (SPADI) which is a valid and reliable index for measuring shoulder pain and disability. It consists of two parts, part one which assesses pain and part two which assesses functional disability. Scores were calculated as follow, in part one pain scores in all questions were added, and the mean value was chosen. In part two functional score of all questions were added and the mean value was chosen for the purpose of data analysis. Final score for each part was statistically analyzed separately.
Range of motion | Baseline
  In this study the shoulder flexion, abduction and internal rotation were measured by using(Model 01129 Guymon goniometer). It is an electrogoniometer which eliminates the need of manually score each measurement by storing the information internally, it reduces time. It measure any joint angle quickly and accurately. It has range of 0 to 360 and stores up to 80 data points. The validity and reliability of electrogoniometer for shoulder assessment was tested and well documented.
Range of motion | 6 weeks
  In this study the shoulder flexion, abduction and internal rotation were measured by using(Model 01129 Guymon goniometer). It is an electrogoniometer which eliminates the need of manually score each measurement by storing the information internally, it reduces time. It measure any joint angle quickly and accurately. It has range of 0 to 360 and stores up to 80 data points. The validity and reliability of electrogoniometer for shoulder assessment was tested and well documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: In one month